CLINICAL TRIAL: NCT06428760
Title: The Effect of Preoperative Subcutaneous Trochanteric Fat Thickness and Trochanteric Soft Tissue Thickness on Postoperative Infection Risk in Patients Undergoing Hemiarthroplasty for Femoral Neck Fracture
Brief Title: Relationship Between Preoperative Subcutaneous Trochanteric Fat Thickness and Postoperative Infection Risk
Status: Not yet recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: ashmehmetonut
Record Dates: First submitted 2024-04-15; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Hip Infection
Keywords: subcutaneous trochanteric fat thickness; infection; femoral neck fracture; soft tissue thickness; obesity; hemiarthroplasty
MeSH Terms: conditions — Infections; Femoral Neck Fractures; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The effect of preoperative subcutaneous trochanteric fat thickness and trochanteric soft tissue thickness on postoperative infection risk in patients undergoing hemiarthroplasty for femoral neck fracture

DETAILED DESCRIPTION:
Obesity is a growing problem for healthcare systems and orthopaedic surgeons, with 29% of the adult population in the UK and 40% in the US affected by obesity. The most commonly used measure of obesity in healthcare is body mass index (BMI), and the World Health Organisation defines obesity as a BMI ≥ 30 kg/m2. Much of the arthroplasty literature has also focused on the use of BMI as a measure of obesity.

BMI-defined obesity is associated with an increased risk of perioperative complications (including infection and dislocation) in total hip arthroplasty. It has also been shown that there is a gradual increase in anaesthetic time, operative time and length of hospital stay as BMI increases in obese patients.

BMI is an imperfect measure because it does not take into account age, sex, race, fat distribution or muscle mass. Previous studies have shown that subcutaneous fat depth (FD) is an independent risk factor for wound infection in cervical and lumbar spine surgery and after laparotomy. It is not known whether increased subcutaneous fat and soft tissue mass are associated with an increased risk of complications after arthroplasty for femoral neck fractures.

The aim of this study was to investigate whether preoperative measurement of subcutaneous adipose tissue by radiography and computed tomography (CT) and muscle thickness in the gluteus medius/minus, gluteus maximus, anterior and medial compartments by computed tomography (CT) in femoral neck fractures correlate with infection rates at postoperative follow-up.

Hypothesis: In patients with high body mass index (BMI) with femoral neck fractures, the investigators believe that the relationship between increased subcutaneous adipose tissue on radiographs and CT sections and wound infection is as effective as the relationship between increased muscle thickness in the gluteus medius/minimus, gluteus maximus, anterior and medial compartments measured on CT sections and wound infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 65 years of age
* Femoral neck fractures
* Female patients
* Patients undergoing hemiarthroplasty

Exclusion Criteria:

* Patients younger than 65 years
* Male patients
* Patients with immunosuppressive conditions
* Intertrochanteric fractures
* Patients with revision surgery
* Pathological femoral neck fractures

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Female patients over 65 years of age who were admitted to our hospital with a history of a femoral neck fracture and who underwent hemiarthroplasty.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-05-30 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Effect of trochanteric fat and soft tissue | Pre-operative
  The aim of this study was to evaluate the effect of peritrochanteric fat thickness and hip soft tissue parameters on postoperative wound infection in patients with femoral neck fracture.
  Peritrochanteric fat thickness will be measured on preoperative radiographs along with sourcil to skin surface, greater trochanter tip to skin surface, and lateral greater trochanter to skin surface values.
  Hip soft tissue assessment will be measured with the parameters of gluteus medius/minus, gluteus maximus, muscle thickness in the anterior and medial compartments on preoperative CT sections.
Wound infection | First 3 months after surgery
  Wound infection is assessed using investigator dressings. In assessing surgical wound infection, an ASEPSIS score will be calculated for each patient to standardise for serous exudate, erythema, purulent exudate, deep tissue separation at the wound site.

SECONDARY OUTCOMES:
Hospital Length of Stay (LOS) | 1 months
  Hospital Length of Stay (LOS): Evaluate the duration of hospitalization following surgery, as prolonged LOS may be associated with increased risk of nosocomial infections including SSIs.
Mortality Rate | 6 months
  Mortality Rate: Assess mortality rates within a defined follow-up period following surgery, as postoperative infections, especially in vulnerable populations such as elderly patients with femoral neck fractures, may contribute to increased mortality.
  Mortality risk is measured by the Charlson comorbidity index.
Body Mass Index | Measured once preoperatively
  It has been suggested that there is a relationship between body mass index and post-operative wound infection. This index is measured in kg/m2 using the patient's height and weight.
Biochemistry Scans | 1 months
  WBC, leukocyte, neutrophil, lymphocyte, albumin, CRP parameters will be evaluated in routine biochemistry scans

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No